CLINICAL TRIAL: NCT04137510
Title: A Prospective, Randomized, Multi-center Study to Assess the Safety of the Orsiro Mission Stent Compared to the Resolute Onyx Stent in Subjects at High Risk for Bleeding in Combination With 1-month Dual Antiplatelet Therapy (DAPT)
Brief Title: Bioflow-DAPT Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biotronik AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C1703; NCT05549440 (obsolete NCT alias)
Record Dates: First submitted 2019-10-22; First posted 2019-10-24 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2023-04

CONDITIONS: Coronary Artery Disease
Keywords: DAPT; Dual antiplatelet therapy; high bleeding risk; HBR; Coronary artery disease; Percutaneous coronary intervention; PCI
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center, international, two-arm randomized controlled clinical study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orsiro (Experimental)
  Interventions: Device: Percutaneous coronary intervention
- Resolute Onyx (Active Comparator)
  Interventions: Device: Percutaneous coronary intervention

INTERVENTIONS:
Device: Percutaneous coronary intervention — It's a non-surgical procedure that uses a catheter to place a stent into a coronary blood vessel in order to open up the vessel.

SUMMARY:
BIOFLOW-DAPT is a prospective, multi-center, international, two-arm randomized controlled clinical study.

A total of 1'948 subjects will be randomized 1:1 to receive either Orsiro Mission or Resolute Onyx. After index procedure, all patients will receive DAPT (ASA + P2Y12 inhibitor) for 30 days, followed by monotherapy with either P2Y12 inhibitor or ASA only until the end of the study.

Clinical follow-up visits will be scheduled at 1, 6 and 12 months post-procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is acceptable candidate for treatment with a DES
2. Subject is considered at high bleeding risk (HBR), defined as meeting one or more of the following criteria at the time of enrollment:

   1. ≥ 75 years of age
   2. Moderate (estimated GFR 30-59 ml/min) or severe (estimated GFR < 30 ml/min) chronic kidney disease or failure (dialysis dependent)
   3. Advanced liver disease, defined as having cirrhosis with or without portal hypertension and with or without gastroesophageal varices.
   4. Cancer (excluding non-melanoma skin cancer) diagnosed or treated within the previous 12 months or actively treated
   5. Anemia with hemoglobin < 11.0 g/dL or requiring transfusion within 4 weeks prior to randomization
   6. Baseline thrombocytopenia defined as a platelet count <100,000/mm3
   7. History of stroke (ischemic or hemorrhagic), previous intracerebral hemorrhage (ICH) (spontaneous at any time or traumatic within the past 12 months) or presence of a brain arteriovenous malformation
   8. History of hospitalization for bleeding within the previous 12 months
   9. Chronic clinically significant bleeding diathesis
   10. Clinical indication for chronic or lifelong oral anticoagulation (OAC) (with a vitamin K antagonist or non-vitamin K OAC)
   11. Clinical indication for chronic or lifelong steroid or oral nonsteroidal anti-inflammatory drug(s) (NSAIDs), other than aspirin
   12. Nondeferrable major surgery on DAPT
   13. Recent major surgery or major trauma within 30 days before PCI
   14. Precise DAPT score ≥ 25
3. Subject is ≥ 18 years or the minimum age required for legal adult consent in the country of enrollment
4. Subject is capable (no legally authorized representative allowed) to provide written informed consent as approved by the Institutional Review Board (IRB)/Ethics Committee (EC) of the respective clinical site prior to any study related procedure
5. Subject is willing to comply with all protocol and follow-up requirements, including agreement to discontinue DAPT at 1 month
6. Subject is eligible for dual antiplatelet therapy treatment with aspirin plus a P2Y12 inhibitor agent for 1-month post index procedure

Exclusion Criteria:

1. Subject who previously experienced a stent or scaffold thrombosis in any coronary vessel
2. Subject has a known allergy to all types of P2Y12 inhibitor (Clopidogrel, Ticagrelor, Prasugrel, Ticlopidine and Cangrelor; thus preventing the use of the appropriate P2Y12 inhibitor), aspirin, both heparin and bivalirudin, L-605 cobalt-chromium (Co-Cr) alloy or one of its major elements (cobalt, chromium, tungsten, nickel), molybdenum, platinum and irridium, silicon carbide, PLLA,polymers, mTOR inhibiting drugs such as zotarolimus or sirolimus, or contrast media
3. Revascularization of any target vessel within 9 months prior to the index procedure or previous PCI of any non-target vessel within 72 hours prior to or during the index procedure
4. 4. Subject with documented left ventricular ejection fraction (LVEF) <30% as evaluated by the most recent imaging exam (i.e. echocardiogram, ventriculogram, MUGA, etc.), but within 90 days pre/procedure or during the index procedure
5. Subject judged by physician as inappropriate for discontinuation from DAPT at 1 month following index procedure, due to another condition requiring chronic DAPT
6. Subject with planned surgery or procedure necessitating discontinuation of P2Y12 inhibitor and/or aspirin within the first month post-index procedure Note - planned staged procedure at the time of index procedure is not allowed
7. Active bleeding at the time of inclusion
8. Subject with a current medical condition with a life expectancy of less than 12 months
9. Subject is currently participating or intends to participate in another investigational drug or device trial within 12 months following the index procedure or any other clinical trial that may interfere with the treatment or protocol of this study
10. Subject is pregnant and/or breastfeeding or intends to become pregnant during the duration of the study
11. In the investigator's opinion, subject will not be able to comply with the follow-up requirements
12. Subjects who need an impartial witness to give an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1948 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Composite of cardiac death, myocardial infarction (MI) and definite or probable stent thrombosis at 12 months | 12 months post-procedure

SECONDARY OUTCOMES:
Rate of definite/probable stent thrombosis according to the ARC definition | until 12 months post-procedure
Rate of MACCE | until 12 months post-procedure
  composite of all-cause death, MI, and stroke
Rate of MACE | until 12 months post-procedure
  composite of cardiac death, MI, and Target Vessel Revascularization (TVR)
Rate of cardiac death or MI | until 12 months post-procedure
  all, target vessel related MI, Q-wave and non Q-wave, ST-related and non ST-related
Rate of all-cause death, cardiac, non-cardiac | until 12 months post-procedure
Rate of stroke, ischemic and hemorrhagic | until 12 months post-procedure
Rate of clinically-indicated TVR | until 12 months post-procedure
Rate of clinically-indicated Target Lesion Revascularization (TLR) | until 12 months post-procedure
Rate of Target Vessel Failure (TVF) | until 12 months post-procedure
  Composite of clinically-driven TVR, cardiac death or target-vessel related MI
Rate of target lesion failure (TLF) | until 12 months post-procedure
  Composite of clinically driven TLR, cardiac death or target vessel related MI
Rate of bleeding according to BARC definition | until 12 months post-procedure
Rate of bleeding according to GUSTO definition | until 12 months post-procedure
Rate of bleeding according to TIMI definition | until 12 months post-procedure
Rate of Device success | until 12 months post-procedure
  Attainment of less than 30% residual stenosis of the target lesion using assigned stent only
Rate of Procedure success | until 12 months post-procedure
  Attainment of less than 30% residual stenosis of the target lesion using assigned stent only without occurrence of in-hospital major adverse cardiac events

CONTACTS AND LOCATIONS:
Overall Officials: Marco Valgimigli, Prof. Dr., Principal Investigator — Cardiocentro Ticino, Via Tesserete 48, 6900 Lugano, Switzerland
Locations (53):
- Australia (3):
  - The Northern Hospital, Epping
  - John Hunter Hospital, New Lambton
  - Royal Perth Hospital, Perth
- Austria (2):
  - Medizinische Universität Graz, Graz
  - Uniklinikum Salzburg, Salzburg
- Belgium (4):
  - AZ St Jan Brugge, Bruges
  - Ziekenhuis Oost Limburg Genk, Genk
  - AZ Delta, Roeselare
  - UCL St Luc, Woluwe-Saint-Lambert
- Denmark (2):
  - Herlev og Gentofte Hospital, Hellerup
  - Roskilde University Hospital, Roskilde
- France (10):
  - CHU Brest, Brest
  - Centre Hospitalier Universitaire de Lille, Lille
  - Hopital Privé Jacques Cartier, Massy
  - CHU Nimes, Nîmes
  - Assistance Publique Hopitaux de Paris (APHP), Paris
  - Assistance Publique Hopitaux de Paris, Paris
  - Clinique Saint Hilaire, Rouen
  - Clinique Pasteur, Toulouse
  - CHU de Toulouse, Toulouse
  - CHRU de Tours, Tours
- Germany (5):
  - Segeberger Kliniken, Bad Segeberg
  - Charite Virchow-Klinikum, Berlin
  - Contilla Herz- und Gefäßzentrum, Elisabeth-Krankenhaus, Essen
  - Klinikum Friedrichshafen GmbH, Friedrichshafen
  - Städtische Kliniken Neuss, Lukaskrankenhaus GmbH, Neuss
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - The Chinese University of Hong Kong, Shatin
- Hungary (3):
  - Semmelweis University, Budapest
  - Somogy County Kaposi Mór Teaching Hospital, Kaposvár
  - University of Pécs, Pécs
- Italy (4):
  - Azienda Ospedaliero - Universitaria Policlinico - Vittorio, Catania
  - Centro Cardiologico Monzino, Milan
  - IRCCS Fondazione Policlinico "San Matteo", Pavia
  - Azienda Ospedaliero-Universitaria, Torrette
- Latvia (2):
  - Sia AK Medical Solutions, Engure
  - Pauls Stradins Clinical University Hospital, Riga
- Institut Jantung Negara, Kuala Lumpur, Malaysia
- Haga Ziekenhuis, The Hague, Netherlands
- Auckland City Hospital, Auckland, New Zealand
- Poland (2):
  - Krakowski Szpital Specjalistyczny im. Jana Pawla, Krakow
  - Miedziowe Centrum Zdrowia, Lubin
- Tan Tock Seng Hospital, Singapore, Singapore
- Spain (3):
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Clinico Universitario de la Valencia, Valencia
  - Hospital Universitario Araba, Vitoria-Gasteiz
- Switzerland (5):
  - Hôpitaux Universitaires de Genève, Geneva
  - Centre Hospitalier Universitaires Vaudoise, Lausanne
  - CardioCentro Ticino, Lugano
  - Hôpital de Morges, Morges
  - Stadtspital Triemli, Zurich
- Thailand (2):
  - Phramongkutklao Hospital, Bangkok
  - Central Chest Institute of Thailand, Bangkok

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Valgimigli M, Wlodarczak A, Tolg R, Merkely B, Kelbaek H, Legutko J, Galli S, Godin M, Toth GG, Lhermusier T, Honton B, Dietrich PL, Stammen F, Ferdinande B, Silvain J, Capodanno D, Cayla G; Bioflow-DAPT Investigators. Biodegradable-Polymer or Durable-Polymer Stents in Patients at High Bleeding Risk: A Randomized, Open-Label Clinical Trial. Circulation. 2023 Sep 26;148(13):989-999. doi: 10.1161/CIRCULATIONAHA.123.065448. Epub 2023 Aug 25. PMID 37624364
- [Derived] Landi A, Wlodarczak A, Tolg R, Kelbaek H, Legutko J, Galli S, Godin M, Toth GG, Lhermusier T, Honton B, Dietrich PL, Stammen F, Ferdinande B, Silvain J, Capodanno D, Cayla G, Valgimigli M; BIOFLOW-DAPT investigators. Design and Rationale of the BIOFLOW-DAPT Trial: a Prospective, Randomized, Multicenter Study to Assess the Safety of the Orsiro Mission Stent Compared to the Resolute Onyx Stent in Subjects at High Risk for Bleeding in Combination with 1-Month Dual Antiplatelet Therapy. J Cardiovasc Transl Res. 2023 Oct;16(5):1135-1143. doi: 10.1007/s12265-023-10400-x. Epub 2023 Jun 1. PMID 37264295
- [Derived] Capodanno D. Another Coronary Stent for Patients at High Bleeding Risk. JACC Cardiovasc Interv. 2021 Sep 13;14(17):1884-1887. doi: 10.1016/j.jcin.2021.07.028. No abstract available. PMID 34503738